CLINICAL TRIAL: NCT04526665
Title: A Double-blind, Randomized, Placebo-Controlled Study and Open-label Long Term Extension to Evaluate the Efficacy and Safety of Elafibranor 80 mg in Patients With Primary Biliary Cholangitis With Inadequate Response or Intolerance to Ursodeoxycholic Acid
Brief Title: Study of Elafibranor in Patients With Primary Biliary Cholangitis (PBC)
Acronym: ELATIVE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505B-319-1; 2019-004941-34 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cholangitis; PBC; Elafibranor
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Intervention Model Description: This is a double-blind (DB), randomized, placebo-controlled study followed by an open-label long term extension (LTE)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Elafibranor 80mg double-blind (Experimental): Study participants will take 1 tablet per day orally before breakfast with a glass of water each morning
  Interventions: Drug: Elafibranor 80mg
- Placebo (Placebo Comparator): Study participants will take 1 tablet per day orally before breakfast with a glass of water each morning
  Interventions: Drug: Placebo
- Elafibranor 80mg open label (Experimental): Study participants will take 1 tablet per day orally before breakfast with a glass of water each morning
  Interventions: Drug: Elafibranor 80mg

INTERVENTIONS:
Drug: Elafibranor 80mg — Elafibranor 80mg daily
  Other Names: Iqirvo®
  Arms: Elafibranor 80mg double-blind; Elafibranor 80mg open label
Drug: Placebo — Placebo daily
  Arms: Placebo

SUMMARY:
The participants of this study will have confirmed Primary Biliary Cholangitis (PBC) with inadequate response or intolerance to ursodeoxycholic acid (which is a medication used in the management and treatment of cholestatic liver disease).

PBC is a slowly progressive disease characterized by damage of the bile ducts in the liver, leading to a buildup of bile acids which causes further damage. The liver damage in PBC may lead to scarring (cirrhosis). PBC may also be associated with multiple symptoms. Many patients with PBC may require liver transplant or may die if the disease progresses and a liver transplant is not done.

The main aim of this study is to determine if elafibranor (the study drug) is better than placebo (a dummy treatment) at decreasing the levels of a specific blood test (alkaline phosphatase) that provides information about participant's disease. This study will also evaluate the safety of long-term treatment with elafibranor, as well as the impact on symptoms such as itchy skin (pruritus) and tiredness (fatigue).

This study has two main parts:

Part 1 will compare a daily dose of elafibranor to a daily dose of placebo and will last between a minimum of one year and a maximum of two years.

Part 2, all participants will receive elafibranor for a period of up to 5 years or until the total treatment duration (part 1 and part 2) reaches 6 years, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

* Males or females age of 18 to 75 years (inclusive)
* Definite or probable Primary biliary cholangitis (PBC) diagnosis
* Alkaline phosphatase (ALP) ≥ 1.67x upper limit of normal (ULN)
* Total bilirubin (TB) ≤ 2x ULN
* Ursodeoxycholic acid (UDCA) for at least 12 months (stable dose ≥ 3 months) prior to screening, or unable to tolerate UDCA treatment (no UDCA for ≥ 3 months) prior to screening (per country standard-of-care dosing)
* Must have PBC Worst Itch Numeric rating scale (NRS) collected prior to randomization
* Females participating in this study must be of non-child bearing potential or must be using highly efficient contraception for the full duration of the study and for 1 month after the last drug intake

Exclusion Criteria:

* History or presence of other concomitant liver disease
* Clinically significant hepatic decompensation, including patients with complications of cirrhosis/portal hypertension
* Medical conditions that may cause non-hepatic increases in ALP (e.g., Paget's disease) or which may diminish life expectancy to < 2 years, including known cancers
* Patient has a positive test for HIV Type 1 or 2 at screening, or patient is known to have tested positive for HIV
* Evidence of any other unstable or untreated clinically significant disease
* History of alcohol abuse
* For female patients: known pregnancy or lactating
* Use of fibrates and glitazones within 2 months prior to screening
* Use of Obeticholic acid (OCA), azathioprine, cyclosporine, methotrexate, mycophenolate, pentoxifylline, budesonide and other systemic corticosteroids (parenteral and oral chronic administration only); potentially hepatotoxic drugs
* (including α-methyl-dopa, sodium valproic acid isoniazid, or nitrofurantoin) within 3 months prior to screening
* Use of antibodies or immunotherapy directed against interleukins (ILs) or other cytokines or chemokines within 12 months prior to screening
* For patients with previous exposure to OCA, OCA should be discontinued 3 months prior to screening
* Patients who are currently participating in, plan to participate in, or have participated in an investigational drug study or medical device study containing active substance within 30 days or five half-lives, whichever is longer, prior to screening; for patients with previous exposure to seladelpar, seladelpar should be discontinued 3 months prior to screening
* Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) values > 5 x ULN
* For patients with AT or TB>ULN at SV1, variability of AT or TB > 40% (see section 3.5.1)
* Albumin<3.0 g/dl
* Severely advanced patients according to Rotterdam criteria (TB > ULN and albumin <LLN)
* INR > 1.3 due to altered hepatic function
* CPK > 2 x ULN
* Screening serum creatinine > 1.5 mg/dl
* Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as patients with markers of kidney failure damage or eGFR < 60 mL/min/1.73 m^2) calculated by Modification of diet in renal disease (MDRD)
* Platelet count < 150 x 10^3/μL
* AFP > 20 ng/mL with 4-phase liver CT or MRI imaging suggesting presence of liver cancer
* Known hypersensitivity to the investigational product or to any of the formulation excipients of the elafibranor or placebo tablet Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2028-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (115):
- United States (46):
  - The Institute for Liver Health, Chandler, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - California Pacific Medical Center - Sutter Pacific Medical Foundation, San Francisco, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - South Denver Gastroenterology, P.C., Englewood, Colorado
  - Yale School of Medicine, Digestive Diseases, New Haven, Connecticut
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Saint Louis University, St Louis, Missouri
  - UPMC Center for Liver Diseases, New Hyde Park, New York
  - NYU Langone Health / NYU Grossman School of Medicine, New York, New York
  - Columbia University Medical Center - Center for Liver Disease and Transplantation, New York, New York
  - The New York-Presbyterian Hospital, David H. Koch Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Centre for Liver disease/ Atrium Health, Huntersville, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Investigational Drug Service Pharmacy Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina- College of Medicine, Charleston, South Carolina
  - Vanderbilt Digestive Disease Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, PLLC, Dallas, Texas
  - The University of Texas Southwestern Medical Center-IDS Aston Pharmacy, Dallas, Texas
  - Texas Digestive Disease Consultants dba GI Alliance, Fort Worth, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - St. Luke's Health-Baylor St Luke's Medical center - Advanced Liver Therapies Research, Houston, Texas
  - American Research Corporation, San Antonio, Texas
  - Gastro health & Nutrition-Victoria, Victoria, Texas
  - Intermountain Medical Center - Transplant Services, Murray, Utah
  - University of Utah Hospital-Division of Gastroenterology, Hepatology, and Nutrition, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Maryview Hospital Inc, Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - Richmond Community Hospital LLC, Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Virginia Commonwealth University Clinical Research Services Unit (CRSU), Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Argentina (6):
  - Hospital Italiano de Buenos Aires, CABA, Buenos Aires
  - Hospital Alemán, Caba, Buenos Aires
  - Hospital Británico de Buenos Aires, CABA, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Espanol De Mendoza, Godoy Cruz, Mendoza Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
- Belgium (4):
  - Hôpital Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospital Leuven, Leuven
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo-HCFMUSP, São Paulo, São Paulo
- Canada (4):
  - University of Calgary Liver Unit - Heritage Medical Research Clinic (HMRC), Calgary, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Division of Gastroenterology, Vancouver, British Columbia
  - Shared Health Inc.-Operating as Health Sciences Centre-John Buhler Research Centre, Winnipeg, Manitoba
  - Centre de Recherche du Centre Hospitalier de l'Université de Montreal (CRCHUM), Montreal
- Chile (5):
  - Hospital de La Serena, La Serena, Coquimbo Region
  - Centro de Investigaciones Clinicas (CIC), Viña del Mar, Región de Valparaíso
  - Clínica Universidad de los Andes, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Centro de Investigacion Clinica Universidad Catolica CICUC, Santiago
- France (10):
  - CHU Amiens Picardie, Amiens
  - Hôpital Henri Mondor, Créteil
  - CHU Grenoble Alpes - Hôpital Albert Michallon, Grenoble
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Hôpital Saint-Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital Haut Lévêque, Pessac
  - Hôpital Robert Debré - CHU de Reims, Reims
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (7):
  - Gastro - Sudien, Berlin
  - Charite - Universitätsmedizin Berlin- CVK - Medizinische Klinik, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Center for Gastroenterology and Hepatology (GHZ) Kiel, Kiel
  - EUGASTRO GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Italy (6):
  - Ospedale Civile di Baggiovara-Struttura Complessa di Medicina ad indririzzo Metabolico Nutrizionale, Modena, Località Baggiovara
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera San Paolo, Dipartimento di Scienza della Salute, UO Medicina VI e Pathologia e Gastroenterologia, Milan
  - ASST Monza - Ospedale San Gerardo, Gastroenterologia, Monza
  - Azienda Ospedale- Università degli Studi di Padova UOC Gastroenterologia, Padua
  - Azienda Ospedaliera Universitaria Policlinico P. Giaccone, UOC di Gastroenterologia-Dip.Medicina Interna e Specialistica, Palermo
- South Africa (3):
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Groote Schuur Hospital, University of Cape Town - Clinical Research Centre, Cape Town, Western Cap
  - Mediclinic Constantiaberg, North Suites, Cape Town
- Spain (9):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro -Madrid, Madrid
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (2):
  - Inselspital, Universitätsspital Bern Universitätsklinik für Viszerale chirurgie und Medizin Hepatologie, Bern
  - Fondazione Epatocentro Ticino, Lugano
- Turkey (Türkiye) (3):
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir, Bornova
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Gastroentoloji Bilim Dali, Istanbul, Pendik
  - Hacette Universitesi Hastenesi IC, Hastaliklari Anabilim Dali, Gastronenteroloji Bilim Dali, Mithapasa Cad. Hacettepe Mah., Ankara
- United Kingdom (8):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust-Freeman Hospital, Newcastle upon Tyne, Newcastle
  - Belfast Health and Social Care Trust-Royal Victoria Hospital, Belfast
  - Frimley Health NHS Foundation Trust - Frimley Park Hospital, Camberley
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge
  - Hull University Teaching Hospitals NHS Trust , Hull Royal Infirmary, Hull
  - King's College Hospital. King's College NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust - Queen's Medical Centre (QMC), Nottingham
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Kowdley KV, Bowlus CL, Levy C, Akarca US, Alvares-da-Silva MR, Andreone P, Arrese M, Corpechot C, Francque SM, Heneghan MA, Invernizzi P, Jones D, Kruger FC, Lawitz E, Mayo MJ, Shiffman ML, Swain MG, Valera JM, Vargas V, Vierling JM, Villamil A, Addy C, Dietrich J, Germain JM, Mazain S, Rafailovic D, Tadde B, Miller B, Shu J, Zein CO, Schattenberg JM; ELATIVE Study Investigators' Group; ELATIVE Study Investigators' Group. Efficacy and Safety of Elafibranor in Primary Biliary Cholangitis. N Engl J Med. 2024 Feb 29;390(9):795-805. doi: 10.1056/NEJMoa2306185. Epub 2023 Nov 13. PMID 37962077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, double-blind (DB), placebo-controlled study followed by an open-label long-term extension (LTE) was conducted in participants with primary biliary cholangitis (PBC) at 82 sites in 14 countries (Argentina, Belgium, Brazil, Canada, Chile, France, Germany, Italy, South Africa, Spain, Switzerland, Turkey, United Kingdom, and United States). First participant was recruited on 24 September 2020 and data cut-off (DCO) date was 01 June 2023.
Pre-assignment Details: This study consisted of a 2- to 12-week screening period, a 52- to 104-week DB period consisting of a 52-week common DB period followed by a variable DB period of up to 52 weeks in duration; a 4- to 5-year LTE period; and a 4-week safety follow-up period after the last dose of study treatment. A total of 161 participants were randomized in 2:1 ratio to receive once daily elafibranor or placebo. Results are presented up to DCO of 01 June 2023.
Groups:
- Elafibranor 80 mg: Participants received elafibranor 80 milligrams (mg) orally once daily before breakfast during the DB period (maximum observed exposure= 104 weeks).
- Placebo: Participants received placebo matched to elafibranor orally once daily before breakfast during the DB period (maximum observed exposure= 106 weeks).
Period: Overall Study
Arm/Group | Elafibranor 80 mg | Placebo
Started | 108 | 53
Completed (Completed DB period) | 94 | 46
Not Completed | 14 | 7
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Death | 2 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Elafibranor 80 mg: Participants received elafibranor 80 mg orally once daily before breakfast during the DB period (maximum observed exposure= 104 weeks).
- Total: Total of all reporting groups
Arm/Group | Elafibranor 80 mg | Placebo | Total
Number analyzed (Participants) | 108 | 53 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (8.4) | 56.4 (9.3) | 57.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 52 | 154
  Male | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 101 | 46 | 147
  Black or African American | 2 | 0 | 2
  Asian | 1 | 3 | 4
  American Indian or Alaska Native | 0 | 1 | 1
  Other | 3 | 2 | 5
  Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Treatment Based on Cholestasis Response at Week 52
Description: Cholestasis response was defined as alkaline phosphatase (ALP) < 1.67 x upper limit of normal (ULN) and total bilirubin (TB) <= ULN and ALP decrease from baseline >= 15% at Week 52 and based on the composite strategy imputing non-response for participants who experienced intercurrent events (ICEs) (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 108 | 53
Percentage of participants | 50.9 [41.6 to 60.2] | 3.8 [1.0 to 12.8]
Statistical Analysis 1: Comparison: Elafibranor 80 mg vs Placebo; Test type: Other; p < 0.0001, Exact Cochran-Mantel-Haenszel test; Exact Cochran-Mantel-Haenszel test stratified by the randomization factors (ALP >3xULN or TB>ULN:Yes/No, and Baseline PBC Worst Itch NRS ≥ 4: Yes/No); Odds Ratio (OR) = 37.562, 95% CI 2-sided [7.641 to 302.247]

2. Secondary Outcome: Key Secondary Endpoint: Percentage of Participants With Response to Treatment Based on ALP Normalization at Week 52
Description: Response to treatment based on normalization of ALP at Week 52 was defined as percentage of participants with ALP =<1.0× ULN and based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 108 | 53
Percentage of participants | 14.8 [9.3 to 22.7] | 0 [0.0 to 6.8]

3. Secondary Outcome: Key Secondary Endpoint: Change From Baseline in Pruritus Based on PBC Worst Itch Numeric Rating Scale (NRS) Score in Participants With Baseline PBC Worst Itch NRS Score ≥4 to Week 52
Description: The PBC Worst Itch NRS is a simple, self-administered patient reported outcome (PRO) questionnaire that measures itch intensity. Participants rate intensity of their worst Itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Total score ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse outcomes. Baseline was defined as the average of the daily PBC Worst itch scores on available data within 14 days prior the day of randomization. Post-baseline data was defined as the average of the daily PBC Worst itch scores on available data in 4-week period intervals (available data every 28 days after the day of first study drug intake).
Time Frame: Baseline (up to 14 days pre-dose) and Week 52
Population: The Pruritus ITT population included all participants from the ITT analysis set with baseline PBC Worst Itch NRS score ≥4. Only those participants with data collected at Week 52 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 44 | 22
Scores on a scale | -1.930 [-2.602 to -1.258] | -1.146 [-2.143 to -0.150]
Statistical Analysis 1: Comparison: Elafibranor 80 mg vs Placebo; Test type: Other; p = 0.1970, mixed model for repeated measures (MMRM); Least square mean difference = -0.784, 95% CI 2-sided [-1.986 to 0.418]

4. Secondary Outcome: Key Secondary Endpoint: Change From Baseline in Pruritus Based on PBC Worst Itch NRS Score in Participants With Baseline PBC Worst Itch NRS Score ≥4 to Week 24
Description: The PBC Worst Itch NRS is a simple, self-administered PRO questionnaire that measures itch intensity. Participants rate intensity of their worst Itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Total score ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse outcomes. Baseline was defined as the average of the daily PBC Worst itch scores on available data within 14 days prior the day of randomization. Post-baseline data was defined as the average of the daily PBC Worst itch scores on available data in 4-week period intervals (available data every 28 days after the day of first study drug intake).
Time Frame: Baseline (up to 14 days pre-dose) and Week 24
Population: The Pruritus ITT population included all participants from the ITT analysis set with baseline PBC Worst Itch NRS score ≥4. Only those participants with data collected at Week 24 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 44 | 22
Scores on a scale | -1.598 [-2.246 to -0.951] | -1.255 [-2.201 to -0.309]
Statistical Analysis 1: Comparison: Elafibranor 80 mg vs Placebo; Test type: Other; p = 0.5522, MMRM; MMRM with treatment, 4-week period and treatment by 4-week period interaction as fixed factors and adjusting for baseline and stratification factors; Least square mean difference = -0.343, 95% CI 2-sided [-1.489 to 0.803]

5. Secondary Outcome: Change From Baseline in ALP at Weeks 4, 13, 26, 39 and 52
Description: Blood samples were collected at specified timepoints for assessment of ALP. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Weeks 4, 13, 26, 39 and 52
Population: The ITT population included all randomized participants. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 104 | 48
Units per Liter (U/L)
  Week 4 | -116.4 (63.1) | -14.3 (92.6)
  Week 13 | -131.8 (74.6) | -19.1 (78.3)
  Week 26: number analyzed (Participants) | 103 | 47
  Week 26 | -126.2 (85.5) | -6.0 (75.6)
  Week 39: number analyzed (Participants) | 99 | 47
  Week 39 | -134.7 (89.8) | -20.0 (90.1)
  Week 52: number analyzed (Participants) | 94 | 47
  Week 52 | -117.7 (96.5) | -8.8 (91.2)

6. Secondary Outcome: Percentage of Participants With ALP Response From Baseline at Week 52
Description: ALP response was defined as ALP decrease from baseline >= 10%; ALP decrease from baseline >= 20% and ALP decrease from baseline >= 40% at Week 52 and based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: The ITT population included all randomized participants. Only those participants with data collected at Week 52 are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 106 | 53
Percentage of participants
  ALP response >= 10% decrease from baseline | 75.5 | 22.6
  ALP response >= 20% decrease from baseline | 69.8 | 5.7
  ALP response >= 40% decrease from baseline | 54.7 | 0.0

7. Secondary Outcome: Percentage of Participants With Response to Treatment According to ALP < 1.5x ULN, ALP Decrease From Baseline >= 40% and TB =<ULN at Week 52
Description: Response to treatment was according to ALP < 1.5x ULN, ALP decrease from baseline >= 40% and TB =<ULN at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 106 | 53
Percentage of participants | 37.7 | 0.0

8. Secondary Outcome: Percentage of Participants With Response to Treatment According to ALP < 3x ULN, Aspartate Aminotransferase (AST) < 2x ULN and TB =< 1 Milligrams Per Deciliter (mg/dL) (Paris I) at Week 52
Description: Response to treatment was according to ALP < 3x ULN, AST < 2x ULN and TB =< 1 mg/dL (Paris I) at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 106 | 53
Percentage of participants | 68.9 | 47.2

9. Secondary Outcome: Percentage of Participants With Response to Treatment According to ALP =< 1.5x ULN, AST =< 1.5x ULN and TB =< 1 mg/dL (Paris II) at Week 52
Description: Response to treatment was according to ALP =< 1.5x ULN, AST =< 1.5x ULN and TB =< 1 mg/dL (Paris II) at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 107 | 53
Percentage of participants | 43.0 | 5.7

10. Secondary Outcome: Percentage of Participants With Response to Treatment According to TB Decrease of 15% Change From Baseline at Week 52
Description: Response to treatment was according to TB decrease of 15% change from baseline at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 105 | 53
Percentage of participants | 31.4 | 22.6

11. Secondary Outcome: Percentage of Participants With Response to Treatment According to Normalization of TB (TB =< ULN) and/or Albumin (ALB >= Lower Limit of Normal [LLN]) (Rotterdam) at Week 52
Description: Response to treatment was according to TB (TB =< ULN) and/or albumin (ALB >= LLN) (Rotterdam) at week 52. Participant was considered as responder at Week 52 only if total bilirubin and albumin were normal. The endpoint was analyzed in participants with abnormal total bilirubin (TB > ULN) or albumin (ALB < LLN) at baseline. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 4 | 2
Percentage of participants
  TB (TB =< ULN) | 25.0 | 50.0
  Albumin (ALB >= LLN): number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Response to Treatment According to TB ≤0.6 x ULN at Week 52
Description: Response to treatment was according to TB ≤0.6 x ULN at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 105 | 53
Percentage of participants | 74.3 | 77.4

13. Secondary Outcome: Percentage of Participants With Response to Treatment According to ALP ≤1.67 x ULN and TB ≤1 mg/dL (Momah/ Lindor) at Week 52
Description: Response to treatment was according to ALP ≤1.67 x ULN and TB ≤1 mg/dL (Momah/ Lindor) at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 106 | 53
Percentage of participants | 51.9 | 9.4

14. Secondary Outcome: Percentage of Participants With Response to Treatment According to no Worsening of TB at Week 52
Description: Response to treatment was according to no worsening of TB, which was defined as level of TB <ULN or no increase from baseline of more than 0.1 x ULN at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 105 | 53
Percentage of participants | 85.7 | 83.0

15. Secondary Outcome: Percentage of Participants With Response to Treatment According to Complete Biochemical Response at Week 52
Description: Response to treatment according to complete biochemical response which was defined as <= ULN values of ALP, TB, AST, ALT and ALB, and international normalized ratio (INR) at Week 52. It was based on the composite strategy imputing non-response for participants who experienced ICEs (study treatment discontinuation or use of rescue therapy for PBC) prior to Week 52.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 107 | 53
Percentage of participants | 9.3 | 0.0

16. Secondary Outcome: PBC 5-, 10- and 15-year Risk Scores Based on United Kingdom (UK)-PBC Score at Week 52
Description: The UK-PBC risk score was defined by the mean percentage risk that a PBC participant treated with UDCA would develop liver failure requiring liver transplantation in 5, 10, and 15 years from diagnosis. It is calculated from the following equation at week 52 as follows: UK-PBC score = 0.0287854*(alpEPxULN-1.722136304) - 0.0422873*([{altastEP x ULN/10}^-1] - 8.675729006) + 1.4199 * (LN(bilEPxULN /10)+2.709607778) - 1.960303*(alb x LLN -1.17673001)-0.4161954*(plt x LLN -1.873564875). The survival S(t) for any given participants was then calculated by S(t) = S0(t) exp(UK-PBC score). Here, alpEP x ULN=ALP /Upper Level Normal ALP at the timepoint, altastEPxULN=(ALT, AST or TA) /upper level normal of the value at the timepoint, bilEP x ULN=bilirubin /upper level normal bilirubin at the timepoint, alb x LLN=alb /alb lower level normal at baseline and plt x LLN=plt/plt lower level normal at baseline. Lower UK-PBC score predicts lower risk and better prognosis.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 93 | 47
Scores on a scale
  UK PBC 5-year risk score | 0.0102 (0.0126) | 0.0146 (0.0264)
  UK PBC 10-year risk score | 0.0330 (0.0393) | 0.0454 (0.0731)
  UK PBC 15-year risk score | 0.0593 (0.0670) | 0.0786 (0.1109)

17. Secondary Outcome: Global PBC Study Group (GLOBE) Score at Week 52
Description: The GLOBE score was a validated risk assessment tool providing an estimate of transplant-free survival for participants with PBC. It was developed by the Global PBC Study Group using Cox regression model on over 4,000 participants with PBC. It is calculated from the following equation at week 52 as follows: GLOBE score = 0.044378 * age at start of ursodeoxycholic acid (UDCA) therapy + 0.93982 * LN (TB x ULN) + 0.335648 * LN (ALP x ULN) - 2.266708 * ALB x LLN - 0.002581 * platelet count per 10^9/L) + 1.216865; where TB x ULN = bilirubin/ULN at the timepoint, ALP x ULN = ALP/ULN at the timepoint, ALB x LLN = ALB/LLN at the timepoint, platelet count per 10^9/L = platelet count per 10^9/L at the timepoint. The Lower GLOBE PBC score predicts lower risk and better prognosis.
Time Frame: At Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 92 | 45
Scores on a scale | -1.03 (0.70) | -0.62 (0.83)

18. Secondary Outcome: Change From Baseline in Hepatobiliary Injury and Liver Function as Assessed by AST, ALT, Gamma-glutamyl Transferase (GGT), 5 Prime Nucleotidase (5'-NT), and Fractionated ALP (Hepatic) (H1 and H2) at Week 52
Description: Hepatobiliary injury and liver function were assessed as measured by AST, ALT, GGT, 5'-NT, and fractionated ALP (hepatic) (H1 and H2). Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: The ITT population included all randomized participants. Only those participants with data collected at Week 52 for each parameter are reported.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 94 | 47
U/L
  AST | -2.5 (17.8) | -4.3 (24.3)
  ALT | -9.7 (22.1) | -6.3 (26.3)
  GGT | -44.0 (95.6) | -17.3 (112.7)
  5'-NT: number analyzed (Participants) | 82 | 43
  5'-NT | -3.63 (5.40) | -2.09 (10.52)
  Hepatic ALP H1: number analyzed (Participants) | 48 | 31
  Hepatic ALP H1 | -107.68 (77.17) | -32.20 (71.42)
  Hepatic ALP H2: number analyzed (Participants) | 48 | 31
  Hepatic ALP H2 | -11.76 (14.67) | -5.20 (54.83)

19. Secondary Outcome: Change From Baseline in Hepatobiliary Injury and Liver Function as Measured by Total and Conjugated Bilirubin at Week 52
Description: Hepatobiliary injury and liver function were assessed as measured by total and conjugated bilirubin. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Micromoles per liter (μmol/L)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 93 | 47
Micromoles per liter (μmol/L)
  Total Bilirubin | -0.67 (3.18) | 0.87 (4.29)
  Conjugated bilirubin: number analyzed (Participants) | 91 | 47
  Conjugated bilirubin | -0.09 (1.98) | 0.61 (2.41)

20. Secondary Outcome: Change From Baseline in Hepatobiliary Injury and Liver Function as Measured by Albumin at Week 52
Description: Hepatobiliary injury and liver function were assessed as measured by albumin. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 94 | 47
Grams per liter (g/L) | 1.0 (2.8) | -1.2 (2.7)

21. Secondary Outcome: Change From Baseline in Hepatobiliary Injury and Liver Function as Measured by INR at Week 52
Description: Hepatobiliary injury and liver function were assessed as measured by INR. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 46
Ratio | 0.028 (0.148) | 0.035 (0.131)

22. Secondary Outcome: Change From Baseline in Biomarkers of Inflammation as Measured by High-sensitivity C-reactive Protein (hsCRP) at Week 52
Description: Biomarkers of inflammation were assessed as measured by hsCRP. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 93 | 47
mg/L | -1.38 (6.53) | 0.22 (2.64)

23. Secondary Outcome: Change From Baseline in Biomarkers of Inflammation as Measured by Fibrinogen and Haptoglobin at Week 52
Description: Biomarkers of inflammation were assessed as measured by fibrinogen and haptoglobin. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 93 | 47
g/L
  Fibrinogen: number analyzed (Participants) | 93 | 46
  Fibrinogen | -1.002 (1.303) | -0.776 (1.265)
  Haptoglobin | -0.185 (0.407) | 0.023 (0.302)

24. Secondary Outcome: Change From Baseline in Biomarkers of Inflammation as Measured by Tumor Necrosis Factor Alpha at Week 52
Description: Biomarkers of inflammation were assessed as measured by TNF-alpha. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 81 | 39
Picograms per milliliter (pg/mL) | -3.346 (15.442) | -0.224 (0.921)

25. Secondary Outcome: Change From Baseline in Immune Response as Measured by Immunoglobulin (Ig)G and IgM at Week 52
Description: Immune response was assessed as measured by IgG and IgM. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 46
g/L
  IgG | -0.423 (1.591) | 0.298 (1.159)
  IgM | -0.606 (0.907) | 0.017 (0.762)

26. Secondary Outcome: Change From Baseline in Biomarkers and Non-invasive Measures of Hepatic Fibrosis as Measured by Enhanced Liver Fibrosis (ELF) and Plasminogen Activator Inhibitor-1 (PAI-1) at Week 52
Description: Biomarkers and non-invasive measures of hepatic fibrosis were assessed as measured by ELF: hyaluronic acid [HA], type 2 procollagen peptide [PIINP], tissue inhibitor of metalloproteinases-1[TIMP-1]) and PAI-1. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Micrograms per liter (mcg/L)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 89 | 44
Micrograms per liter (mcg/L)
  HA | 7.93 (80.35) | 16.36 (48.60)
  PIINP: number analyzed (Participants) | 81 | 32
  PIINP | -2.79 (32.55) | -5.60 (20.03)
  TIMP-1 | -3.03 (51.06) | 23.26 (65.03)
  PAI-1: number analyzed (Participants) | 80 | 40
  PAI-1 | 0.053 (3.032) | 0.785 (7.028)

27. Secondary Outcome: Change From Baseline in Biomarkers and Non-invasive Measures of Hepatic Fibrosis as Measured by Cytokeratin-18 (CK-18) at Week 52
Description: Biomarkers and non-invasive measures of hepatic fibrosis were assessed as measured by CK-18 (M30 and M65). Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 83 | 42
Picomoles per liter (pmol/L)
  CK-18 M30 | -70.71 (444.31) | -5.39 (334.22)
  CK-18 M65: number analyzed (Participants) | 46 | 23
  CK-18 M65 | -50.02 (246.28) | -83.73 (481.30)

28. Secondary Outcome: Change From Baseline in Biomarkers and Non-invasive Measures of Hepatic Fibrosis as Measured by Transforming Growth Factor Beta (TGF-beta) at Week 52
Description: Biomarkers and non-invasive measures of hepatic fibrosis were assessed as measured by TGF-beta. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 8 | 6
pg/mL | 713.074 (6553.956) | -6172.360 (3279.127)

29. Secondary Outcome: Change From Baseline in Liver Stiffness Measured by Transient Elastography (TE) at Week 52
Description: FibroScan® TE device (Echosens, Paris, France) is a non-invasive technique used to measure liver stiffness, which correlated with fibrosis. Baseline was defined as the last non-missing value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilopascal (kPa)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 90 | 44
Kilopascal (kPa) | -0.16 (3.70) | 0.35 (6.39)

30. Secondary Outcome: Change From Baseline in Lipid Parameters at Week 52
Description: Blood samples were collected at specified timepoints for assessment of total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, very low-density lipoprotein (VLDL) cholesterol and triglycerides (TG). Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 47
Millimoles per liter (mmol/L)
  Total cholesterol: number analyzed (Participants) | 94 | 47
  Total cholesterol | -0.532 (0.910) | -0.318 (1.144)
  LDL cholesterol: number analyzed (Participants) | 91 | 47
  LDL cholesterol | -0.428 (0.730) | -0.274 (1.086)
  HDL cholesterol | 0.011 (0.364) | -0.056 (0.399)
  VLDL cholesterol: number analyzed (Participants) | 91 | 47
  VLDL cholesterol | -0.118 (0.159) | 0.015 (0.156)
  TG: number analyzed (Participants) | 92 | 47
  TG | -0.268 (0.370) | 0.031 (0.343)

31. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: Blood samples were collected at specified timepoints for assessment of FPG. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 90 | 42
mmol/L | -0.267 (0.861) | 0.086 (0.381)

32. Secondary Outcome: Change From Baseline in Bile Acids and Biomarkers of Bile Acid Synthesis at Week 52
Description: Blood samples were collected at specified timepoints for assessment bile acids and biomarkers of bile acid synthesis. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 65 | 38
µmol/L
  Chenodeoxycholic acid | 0.177 (0.807) | 0.100 (0.527)
  Cholic acid | 0.156 (0.656) | 0.027 (0.337)
  Deoxycholic acid | -0.027 (0.288) | -0.039 (0.360)
  Glycochenodeoxycholic acid | -0.564 (3.310) | 0.581 (4.408)
  Glycocholic acid | -0.370 (2.422) | 2.253 (12.291)
  Glycodeoxycholic acid | -0.516 (1.247) | -0.266 (2.688)
  Glycolithocholic acid | -0.0234 (0.0762) | -0.0187 (0.1768)
  Lithocholic acid | -0.010 (0.047) | -0.003 (0.047)
  Taurochenodeoxycholic acid | -0.085 (2.495) | 0.857 (3.048)
  Taurocholic acid | 0.070 (2.059) | 1.127 (4.380)
  Taurodeoxycholic acid | -0.0828 (0.4412) | -0.0343 (0.3683)
  Taurolithocholic acid | -0.0098 (0.0424) | -0.0082 (0.0684)

33. Secondary Outcome: Change From Baseline at Week 52 in Bile Acids and Biomarkers of Bile Acid Synthesis as Measured by 7 Alpha-hydroxy-4-cholesten-3-one (C4) at Week 52
Description: Blood samples were collected at specified timepoints for assessment of bile acids and biomarkers of bile acid synthesis as measured by C4. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 61 | 30
mcg/L | -7.288 (16.779) | -4.044 (12.995)

34. Secondary Outcome: Change From Baseline in Bile Acids and Biomarkers of Bile Acid Synthesis as Measured Fibroblast Growth Factor 19 at Week 52
Description: Blood samples were collected at specified timepoints for assessment bile acids and biomarkers of bile acid synthesis as measured by Fibroblast Growth Factor 19. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 73 | 36
pg/mL | -12.89 (80.24) | 54.54 (343.47)

35. Secondary Outcome: Percentage of Participants With Response in PBC Worst Itch NRS Score at Weeks 24 and 52
Description: The PBC Worst Itch NRS is a simple, self-administered PRO questionnaire that measures itch intensity. Participants rate intensity of their worst Itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Total score ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse outcomes. Response to PBC Worst Itch NRS was according to clinically meaningful change at least 30% reduction; one point, two points or three points decrease in score from baseline in participants with a baseline NRS score ≥4. Baseline was defined as the average of the daily PBC Worst itch scores on available data within 14 days prior the day of randomization. Post-baseline data was defined as the average of the daily PBC Worst itch scores on available data in 4-week period intervals (available data every 28 days after the day of first study drug intake).
Time Frame: Baseline (up to 14 days pre-dose) and at Week 24 and Week 52
Population: The Pruritus ITT population included all participants from the ITT analysis set with baseline PBC Worst Itch NRS score ≥4. Only those participants with data collected at Weeks 24 and 52 are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 39 | 21
Percentage of participants
  Week 24: 30% reduction from baseline | 43.6 | 28.6
  Week 52: 30% reduction from baseline: number analyzed (Participants) | 36 | 18
  Week 52: 30% reduction from baseline | 55.6 | 33.3
  Week 24: One-point decrease from baseline | 53.8 | 42.9
  Week 52: One-point decrease from baseline: number analyzed (Participants) | 36 | 18
  Week 52: One-point decrease from baseline | 61.1 | 38.9
  Week 24: Two-point decrease from baseline | 38.5 | 28.6
  Week 52: Two-point decrease from baseline: number analyzed (Participants) | 36 | 18
  Week 52: Two-point decrease from baseline | 47.2 | 33.3
  Week 24: Three-point decrease from baseline | 28.2 | 19.0
  Week 52: Three-point decrease from baseline: number analyzed (Participants) | 36 | 18
  Week 52: Three-point decrease from baseline | 41.7 | 33.3

36. Secondary Outcome: Percentage of Participants With no Worsening of Pruritus as Measured by the PBC Worst Itch NRS Score at Weeks 24 and 52
Description: The PBC Worst Itch NRS is a simple, self-administered PRO questionnaire that measures itch intensity. Participants rate intensity of their worst Itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Total score ranged from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicated worse outcomes. Baseline was defined as the average of the daily PBC Worst itch scores on available data within 14 days prior the day of randomization. Post-baseline data was defined as the average of the daily PBC Worst itch scores on available data in 4-week period intervals (available data every 28 days after the day of first study drug intake). A worsening of Pruritus was defined by a positive change from baseline in PBC Worst Itch NRS score greater than 2 at week 24 and 52.
Time Frame: Baseline (up to 14 days pre-dose) and at Week 24 and Week 54
Population: The Pruritus ITT population included all participants from the ITT analysis set with baseline PBC Worst Itch NRS score ≥4.. Only those participants with data collected at Week 24 and Week 54 are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 93 | 51
Percentage of participants
  Week 24 | 89.2 | 86.3
  Week 52: number analyzed (Participants) | 90 | 46
  Week 52 | 76.7 | 82.6

37. Secondary Outcome: Change From Baseline in 5-D Itch at Week 52
Description: The 5-D Itch scale is a questionnaire that has been validated in several different diseases. It assesses symptoms in terms of 5 domains: duration: score range 1 (less than 6 hours) to 5 (all day); degree: score range 1 (not present) to 5 (unbearable); duration: score range 1 (less than 6 hours) and 5 (all day); direction: score range 1(completely resolved) and 5 (getting worse); disability: score range 1 (never affects or not applicable) and 5 (delays falling asleep and frequently wakes up at night or always affects this activity) and distribution: where the question was to mark where itching is present in body parts over the last two weeks. Participants rated their symptoms over preceding 2-week period on a 1 to 5 scale, with 5 being the most affected. The 5-D Itch total score ranged between 5 (no pruritus) and 25 (most severe pruritus). Higher scores indicated worse outcomes. Baseline= last non-missing value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 46
Scores on a scale | -1.9 [-2.6 to -1.3] | -0.6 [-1.6 to 0.3]

38. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7a at Week 52
Description: The PROMIS Fatigue Short Form 7a consists of seven items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week. Participants completed the PROMIS Fatigue Short Form 7a and answered following questions on a scale from 1 (never) to 5 (always) : "How often did you feel tired"; "How often did you experience extreme exhaustion"; "How often did you run out of energy"; "How often did your fatigue limit you at work"; "How often were you too tired to think clearly"; "How often were you too tired to take a bath or shower" and 'How often did you have enough energy to exercise strenuously". T-score values include mean of 50 and standard deviation of 10. The PROMIS Fatigue T-score ranged from 29.4 (best) to 83.2 (worst). Higher scores indicated worse outcomes. Baseline was defined as the last non-missing value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 46
T-score | -2.45 [-3.84 to -1.07] | -1.23 [-3.22 to 0.77]

39. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) at Week 52
Description: The ESS is a short, self-administered questionnaire that consists of 8 questions asking to rate how likely it is to fall asleep in everyday situations (each question can be scored from 0 to 3 points; '0' indicates no chance of dozing and '3' indicates high chance of dozing). It provides a total score which has been shown to relate to the participant's level of daytime sleepiness (total score range 0 [no sleepiness] to 24 points [significant sleepiness]). The total score is the sum of all item scores and ranged from 0 (best) to 24 (worst). Higher scores indicated more chances of sleepiness. Participants were asked to complete the ESS with regard to the level of sleepiness they experienced over approximately the past 7 days. Baseline was defined as the last non-missing value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 46
Scores on a scale | -0.3 [-1.1 to 0.5] | -0.5 [-1.7 to 0.6]

40. Secondary Outcome: Change From Baseline in PBC-40 at Week 52
Description: PBC-40 assess symptoms across 6 domains:symptoms,itch,fatigue,cognitive,emotional and social. Participants responded on verbal response scale,depending on section options range from 'never'/'not at all'/'strongly disagree' to 'always'/'very much'/'strongly agree'.5 items (3/3 in itch domain and 2/10 in social domain)also included a 'does not apply' option.Domains:Symptoms(7 questions)score range 7-35,Itch(3 questions)score range 3-15,Fatigue(11 questions)score range 11-55,Cognitive(6 questions)score range 6-30,Emotional(3 questions)score range 3-15,Social(10 questions)score range 10-50.Score for each domain was provided(total score was not calculated),with each verbal response scale correlating to score of 1-5 per item(0-5 on items with a 'does not apply' option);5=most affected.Individual item scores are summed to give total domain score.Higher scores=worse outcomes.PBC-40 had 4-week recall period.Baseline=last non-missing value on or before first dose of randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 95 | 46
Scores on a scale
  Symptoms | 0.2 [-0.5 to 0.8] | -0.9 [-1.8 to 0.1]
  Itch | -1.4 [-1.8 to -0.9] | -0.2 [-0.9 to 0.5]
  Fatigue | -1.5 [-2.7 to -0.2] | -1.2 [-3.0 to 0.7]
  Cognitive | -0.6 [-1.4 to 0.2] | -0.7 [-1.8 to 0.4]
  Emotional | -0.8 [-1.2 to -0.3] | -0.6 [-1.2 to 0.1]
  Social | -1.1 [-2.3 to 0.1] | -0.4 [-2.1 to 1.3]

41. Secondary Outcome: Change From Baseline in Health Utility as Measured by the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) at Week 52
Description: The EQ-5D-5L is a 6-item, standardized questionnaire that assesses mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and overall health state. The visual analog scale (VAS) of EQ-5D-5L questionnaire is numbered from 0 (worst) to 100 (best). Higher scores indicated better outcomes. Baseline was defined as the last non-missing value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 94 | 46
Scores on a scale | 2.5 [0.0 to 4.9] | 1.6 [-1.9 to 5.0]

42. Secondary Outcome: Change From Baseline in T-Scores for Bone Mineral Density Assessed by Dual-energy X-ray Absorptiometry (DEXA) Scanning at Week 52
Description: DEXA scanning (hip and lumbar) was performed in participants to assess bone mineral density (femoral neck, lumbar and total hip). T-scores were calculated based on actual measured bone density value. The T-score compared a participant's bone density against that of a healthy 30-year-old adult. T-scores were used to determine primary osteoporosis, which exists on its own without any other cause and were divided into 3 categories: low risk, medium risk, and high risk (osteoporosis). T-scores measure the number of minerals in a participant's bone. A participant's level of bone loss was compared to that of a typical, healthy 30-year-old adult. A score ≥-1.0 indicates low risk, medium risk is a score between-2.5 and -1.0, and a high risk/osteoporosis is a score ≤-2.5. A positive change in T-score indicates an improvement in bone mineral density. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 64 | 27
T-score
  Femoral Neck Bone Mineral Density T-score: number analyzed (Participants) | 63 | 27
  Femoral Neck Bone Mineral Density T-score | -0.016 (0.402) | -0.111 (0.533)
  Lumbar Bone Mineral Density T-score: number analyzed (Participants) | 64 | 26
  Lumbar Bone Mineral Density T-score | -0.006 (0.487) | -0.022 (0.405)
  Total Hip Bone Mineral Density T-score: number analyzed (Participants) | 59 | 24
  Total Hip Bone Mineral Density T-score | 0.039 (0.529) | -0.371 (0.618)

43. Secondary Outcome: Change From Baseline in Serum Markers of Bone Turnover Carboxy Terminal Crosslinked Telopeptides of Type 1 Collagen [CTX] at Week 52
Description: Blood samples were collected at specified timepoints for assessment of serum markers of bone turnover, CTX. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 81 | 32
pg/mL | 36.5 (212.6) | 44.5 (129.7)

44. Secondary Outcome: Change From Baseline in Serum Markers of Bone Turnover Type 1 Procollagen Peptide [P1NP]) at Week 52
Description: Blood samples were collected at specified timepoints for assessment of serum markers of bone turnover, P1NP. Baseline was defined as the last non-missing central value on or before the first dose of the randomized study medication.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 81 | 32
mcg/L | -2.79 (32.55) | -5.60 (20.03)

45. Secondary Outcome: Percentage of Participants With Onset of Clinical Outcomes
Description: Onset of clinical outcomes were described as a composite endpoint composed of the following: model for end stage liver disease sodium (MELD-Na) >14 for participants with baseline MELD-Na <12; liver transplant; uncontrolled ascites requiring treatment; hospitalization for new onset or recurrence of any including, variceal bleed, hepatic encephalopathy defined as West-Haven score of 2 or more and spontaneous bacterial peritonitis; and death.
Time Frame: From Day 1 up to Week 52
Population: The ITT population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 108 | 53
Percentage of participants
  Meld-Na > 14 while baseline Meld-Na < 12 | 0.9 | 0.0
  Liver transplant | 0.0 | 0.0
  Uncontrolled ascites requiring treatment | 0.9 | 0.0
  Hospitalization for new onset or recurrence of variceal bleed | 0.0 | 0.0
  Hospitalization for new onset or recurrence of Hepatic encephalopathy | 0.0 | 0.0
  Hospitalization for new onset or recurrence of Spontaneous bacterial peritonitis | 0.0 | 0.0
  Death | 0.9 | 0.0

46. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant who was administered an investigational product, and which does not necessarily have a causal relationship with treatment. A TEAE was defined as any AE with onset during TEAE assessment period, or any event started prior to first dose of treatment and worsened or became serious during the TEAE assessment period. An SAE was any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality/birth defect. An AESI was an AE that might not be serious but was of special importance to a particular treatment or class.
Time Frame: TEAEs were collected from the start of study treatment administration (Day 1) up to DCO date of 01 June 2023, approximately 980 days.
Population: Safety analysis set included all participants who were administered at least one dose of DB study drug irrespective of the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Placebo
Number analyzed (Participants) | 108 | 53
Participants
  TEAEs | 104 | 48
  TESAEs | 11 | 7
  AESIs | 32 | 14

47. Secondary Outcome: Plasma Concentrations of Elafibranor and GFT1007
Description: Blood samples were collected at specified timepoints to evaluate plasma concentration of Elafibranor and its metabolite GFT1007.
Time Frame: Week 4: pre-dose, 0.5 hour, 1.5 hours, between 2-3 hours, 4 hours and 6 hours post-dose
Population: Pharmacokinetics Analysis Set included all participants who were administered at least one dose of elafibranor and have at least one post-dose PK sample. Only those participants with data collected at specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Elafibranor 80 mg
Number analyzed (Participants) | 103
Nanograms per milliliter (ng/mL)
  Elafibranor: Week 4: Pre-dose: number analyzed (Participants) | 100
  Elafibranor: Week 4: Pre-dose | 92.7 (52.9)
  Elafibranor: Week 4: 0.5 hour post-dose | 408.2 (104.1)
  Elafibranor: Week 4: 1.5 hours post-dose: number analyzed (Participants) | 102
  Elafibranor: Week 4: 1.5 hours post-dose | 281.7 (66.1)
  Elafibranor: Week 4: between 2-3 hours post-dose | 182.0 (67.8)
  Elafibranor: Week 4: 4 hours post-dose: number analyzed (Participants) | 101
  Elafibranor: Week 4: 4 hours post-dose | 127.7 (52.7)
  Elafibranor: Week 4: 6 hours post-dose: number analyzed (Participants) | 101
  Elafibranor: Week 4: 6 hours post-dose | 117.1 (53.5)
  GFT1007: Week 4: Pre-dose: number analyzed (Participants) | 100
  GFT1007: Week 4: Pre-dose | 77.3 (85.6)
  GFT1007: Week 4: 0.5 hour post-dose: number analyzed (Participants) | 102
  GFT1007: Week 4: 0.5 hour post-dose | 894.6 (150.0)
  GFT1007: Week 4: 1.5 hours post-dose: number analyzed (Participants) | 102
  GFT1007: Week 4: 1.5 hours post-dose | 1707.2 (52.1)
  GFT1007: Week 4: between 2-3 hours post-dose | 1160.8 (53.9)
  GFT1007: Week 4: 4 hours post-dose: number analyzed (Participants) | 101
  GFT1007: Week 4: 4 hours post-dose | 655.8 (54.7)
  GFT1007: Week 4: 6 hours post-dose: number analyzed (Participants) | 101
  GFT1007: Week 4: 6 hours post-dose | 375.7 (65.9)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were reported from the start of study treatment administration (Day 1) up to DCO date of 01 June 2023, approximately 980 days.
Description: Safety analysis set included all participants who were administered at least one dose of DB study drug irrespective of the treatment received.
Arm/Group | Elafibranor 80 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/108 | 0/53
Serious Adverse Events (participants affected / at risk) | 11/108 | 7/53
Other Adverse Events (participants affected / at risk) | 103/108 | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elafibranor 80 mg (N=108) | Placebo (N=53)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elafibranor 80 mg (N=108) | Placebo (N=53)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10) | 3 (5)
Constipation (Gastrointestinal disorders) | 9 (11) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (13) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (13) | 3 (3)
Vomiting (Gastrointestinal disorders) | 12 (15) | 1 (1)
Fatigue (General disorders) | 10 (10) | 7 (8)
Pain (General disorders) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 31 (31) | 19 (19)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 12 (16) | 9 (10)
Abnormal weight gain (Metabolism and nutrition disorders) | 21 (21) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (4)
Headache (Nervous system disorders) | 9 (9) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (26) | 14 (14)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT04526665/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04526665/SAP_001.pdf